CLINICAL TRIAL: NCT02083822
Title: Cerebral Abnormalities Detected by MRI, Realized at the Age of Term and the Emergence of Executive Functions
Acronym: EPIRMEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRN11-ES / EPIRMEX
Record Dates: First submitted 2013-12-13; First posted 2014-03-11 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Premature Baby 25 to 32 Weeks
Keywords: premature baby; MRI : conventional and advanced images; Executive function testing at 5 years of age
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI assessment (Experimental)
  Interventions: Procedure: term MRI, executive EF functions testing

INTERVENTIONS:
Procedure: term MRI, executive EF functions testing — An MRI will be realized at term born between 25 and 32 weeks GA

SUMMARY:
The survival of premature babies increased during the last decades. However, the neurocognitive long term development of these children is worrying, as demonstrated by EPIPAGE 1 study.

These children present high risk of deficits such as cognitive deficits, adaptive malfunction, behavior disorders and difficulties in school learning.

Understanding the specific neuropsychological disorders at the origin of these deficits is an important objective. Studies realized at school age showed that many premature children have executive functions (EF) disorders. However the specific nature of these disorders and the neuropathology associated are unknown.

The aim of this study is to realise MRI at term age in preterm babies born less than 32 GA and to correlate MRI findings with executives functions and neurodevelopmental outcome

DETAILED DESCRIPTION:
An MRI would be realized between 39 and 41 GA

At the age of 5 years, executive functions and neurodevelopmental testing would be realized.

600 newborns were recruited.

ELIGIBILITY:
Inclusion Criteria

Infants who were :

* born between 25 and 32 WGA
* hospitalized in a neonatology service which participate to the present study
* included in EPIPAGE 2 follow-up study
* infants whose parents had signed the consent agreement and benefit from national health insurance

Exclusion Criteria

* Infants with congenital abnormalities

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2011-06; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Executive functions evaluation at age of 5 and comparison with conventionnal and advanced MRI imagings | During the 5 years follow up

SECONDARY OUTCOMES:
Perinatal risk factors and cerebral lesions as assessed on MRI | During the 5 years follow up
Perinatal risk factors and executive and cognitive functions evaluated at 5 years of age | During the 5 years follow up

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Service de Neurologie Pédiatrique, Angers
  - Service de Néonatologie, Bordeaux
  - Service de Néonatologie, Caen
  - Médecine Néonatale et Réanimation Pédiatrique, Grenoble
  - Service de REANIMATION NEONATALE ET PEDIATRIQUE, NEONATOLOGIE, Le Kremlin-Bicêtre
  - Service de Néonatologie, Lille
  - Médecine Infantile - Néonatologie - Périnatologie, Marseille
  - Service de Néonatalogie, Marseille
  - Service de Néonatologie, Nancy
  - Service de Néonatologie, Nantes
  - Réanimation néonatale et Néonatologie, Paris
  - Service de Réanimation, Néonatologie, Reims
  - Service de Néonatologie, Rennes
  - Service de Pédiatrie Néonatale et Réanimation, Rouen
  - Service de Réanimation pédiatrique, Néonatologie, Tours